CLINICAL TRIAL: NCT04167358
Title: Long-term Safety and Tolerability Study of Linerixibat for the Treatment of Cholestatic Pruritus in Participants With Primary Biliary Cholangitis
Brief Title: Linerixibat Long-term Safety, and Tolerability Study
Acronym: LLSAT
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 212358; 2019-003158-10 (EudraCT Number)
Expanded Access: NCT05448170 (Available)
Record Dates: First submitted 2019-11-15; First posted 2019-11-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Cholestasis
Keywords: Linerixibat; Cholestasis; Cholestatic pruritus; Primary biliary cholangitis; LLSAT
MeSH Terms: conditions — Cholestasis; Liver Cirrhosis, Biliary

STUDY DESIGN:
Intervention Model Description: This is a non-comparator single group study.
Masking Description: This is an open label non-comparator study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants receiving linerixibat (Experimental): Participants who previously participated in the Phase 2 studies (BAT117213 and 201000 GLIMMER [Group 1]) and Phase 3 study (212620 GLISTEN [Group 2]), will receive linerixibat.
  Interventions: Drug: Linerixibat

INTERVENTIONS:
Drug: Linerixibat — All participants will receive linerixibat.

SUMMARY:
This is an open-label, non-comparator, global, multi-center, long-term safety study for evaluating safety and tolerability of linerixibat in participants with cholestatic pruritus in primary biliary cholangitis (PBC) who participated in a prior clinical trial with linerixibat (BAT117123 [NCT01899703], 201000 GLIMMER [NCT02966834] (group 1) or 212620 GLISTEN [NCT00210418]) (group 2). All participants will receive open-label linerixibat for the duration of the study. The study duration is expected to last until the study's end or until linerixibat can be lawfully made available to participants. However, the total duration of study participation will vary by participant depending upon the time of entry relative to study end in their respective country.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants must be 18 to 80 years of age inclusive, at the time of signing the informed consent in the participant's parent trial BAT117213, GLIMMER or GLISTEN.
* Participants with a diagnosis of PBC and a history of associated pruritus as evidenced by randomization into a prior eligible linerixibat clinical trial (BAT117213, GLIMMER or GLISTEN).
* Participants must have completed the main treatment period in a prior eligible linerixibat clinical trial (BAT117213, GLIMMER or GLISTEN).
* A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies: a) is a woman of non-childbearing potential (WONCBP) or b) is a woman of childbearing potential (WOCBP) and using an acceptable contraceptive method.
* Capable of giving signed informed consent.

Exclusion Criteria:

* Screening total bilirubin >2x upper limit of normal (ULN).
* Screening alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >6x ULN.
* Screening estimated glomerular filtration rate (eGFR) <30 milliliters per minute per 1.73 square meter (mL/min/1.73m^2) based on the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation.
* Presence of hepatic decompensation (e.g., variceal bleeds, encephalopathy or ascites).
* Presence of actively replicating viral hepatitis B or C (Viral Hepatitis B [HBV], viral Hepatitis C [HCV]) infection), primary sclerosing cholangitis (PSC), alcoholic liver disease and/or confirmed hepatocellular carcinoma or biliary cancer.
* Current clinically significant diarrhea in the Investigator's medical opinion.
* Current symptomatic cholelithiasis or cholecystitis.
* Current diagnosis or previous diagnosis of colorectal cancer.
* Any current malignancies (including hematologic and solid malignancies).
* History of bariatric surgery with ileal bypass at any time, or any bariatric surgery performed in the past 3 years.
* Use of Obeticholic acid: within 8 weeks prior to the date of the screening visit and may not restart until after the end of the study or early study withdrawal.
* Administration of any other ileal bile acid transporter (IBAT) inhibitor in the 1 month prior to screening until after the end of the study or early study withdrawal.
* QT interval corrected (QTc) >480 millisecond (msec) at screening (12-lead ECG)
* Participants with moderate (or greater) alcohol consumption defined as more than one standard drink per day for women and two drinks per day for men.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2020-07-14 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with non-serious adverse events (AEs) and Serious AEs (SAEs) | Up to 66 months
  AEs and SAEs will be collected.
Number of participants with Severe AEs | Up to 66 months
  AEs and SAEs will be collected.

SECONDARY OUTCOMES:
Change in domain scores of the PBC-40 over time | Baseline and up to 65 months
  The PBC-40 is a participant-derived, disease specific health-related quality of life (QoL) measure with data to support its validity in PBC. The PBC-40 measure is comprised of 40 questions, each scored on a scale of 1 to 5 (where 1 = least impact, 5 = greatest impact) grouped into six domains (symptoms, itch, fatigue, cognition, social, and emotional).
Change in health-related quality of life (QoL) by the Euro Quality-5 dimension-3 level (EQ-5D-3L) scores over time (Group 1 only) | Baseline and up to 65 months
  The EQ-5D-3L is a standardized instrument developed by the EuroQol Group as a measure of health-related quality of life that can be used in a wide range of health conditions and treatments. The EQ-5D consists of a descriptive system and the EQ Visual Analogue Scale (VAS). The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: 1=no problems, 2=some problems, and 3=extreme problems.
Change in self-rated health by EQ VAS scores over time (Group 1 only) | Baseline and up to 65 months
  The EQ-5D-3L is a standardized instrument developed by the EuroQol Group as a measure of health-related quality of life that can be used in a wide range of health conditions and treatments. The EQ-5D consists of a descriptive system and the EQ VAS. The EQ VAS records self-rated health on a vertical visual analogue scale where the endpoints are labelled 'Best imaginable health state' and 'Worst imaginable health state'.
Change in the Beck Depression Inventory (BDI-II) scores over time | Baseline and up to 65 months
  The BDI-II is a 21-item questionnaire used to assess the intensity of depression in clinical and normal participants. Each item is scored from 0 (Normal) to 3 (Severe). The total score on the BDI-II ranges from 0-63, with higher scores reflecting higher levels of depression.
Number of participants with clinically significant changes in hematology, biochemistry (including lipid and liver parameters), and coagulation parameters | Baseline and up to 65 months
  Blood samples will be collected for the analysis of hematology, biochemistry (including lipid and liver parameters) and coagulation parameters.
Percentage of responders at Week 24 and Week 52 of continuous treatment (Group 2 only) | Week 24 and Week 52 of continuous treatment
  Monthly Itch Score (MIS) will be assessed using an numerical rating scale (NRS), ranging from 0 to 10, where 0 represents no itching and 10 the worst imaginable itching. Response thresholds of greater than or equal to (>=) 2, >=3, and >=4-point reduction in MIS will be assessed.
Percentage of participants with maintenance of efficacy at Week 52 of continuous treatment in those that were responders at Week 24 of continuous treatment (Group 2 only) | Week 52 of continuous treatment
  The MIS will be assessed using an NRS, ranging from 0 to 10, where 0 represents no itching and 10 the worst imaginable itching. Maintenance of efficacy occurs when a participant is a responder (>=2, >=3, and >=4-point reduction in MIS) at Week 24 of continuous treatment and is also a responder at Week 52 of continuous treatment.
Change from Baseline Monthly Sleep Score (MSS) (Group 2 only) | Baseline and up to Week 52 of continuous treatment
  The MSS will be assessed using an NRS, ranging from 0 to 10, where 0 represents no sleep interference and 10 is complete sleep interference. This will be assessed at Week 52 of continuous treatment.
Change from Baseline in Monthly Fatigue Score (MFS)(Group 2 only) | Baseline and up to Week 52 of continuous treatment
  The MFS will be assessed using an NRS, ranging from 0 to 10, where 0 represents no fatigue and 10 the worst possible fatigue. This will be assessed at Week 52 of continuous treatment.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (87):
- United States (11):
  - GSK Investigational Site, Davis, California
  - GSK Investigational Site, West Hollywood, California
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Morrisville, North Carolina
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Seattle, Washington
- Argentina (6):
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Capital Federal
  - GSK Investigational Site, Ciudad AutOnoma de Buenos Aire
  - GSK Investigational Site, Ciudad Autonoma de Bueno
  - GSK Investigational Site, Rosario
  - GSK Investigational Site, Santa Fe
- Brazil (4):
  - GSK Investigational Site, Porto Alegre, Rio Grande do Sul
  - GSK Investigational Site, Botucatu
  - GSK Investigational Site, Brasília
  - GSK Investigational Site, Salvador
- GSK Investigational Site, Sofia, Bulgaria
- Canada (2):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Toronto, Ontario
- China (8):
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Changchun
  - GSK Investigational Site, Chongqing
  - GSK Investigational Site, Guangzhou
  - GSK Investigational Site, Nanchang
  - GSK Investigational Site, Nanjing
  - GSK Investigational Site, Shanghai
  - GSK Investigational Site, Tianjin
- Czechia (2):
  - GSK Investigational Site, Pilsen
  - GSK Investigational Site, Prague
- GSK Investigational Site, Lille, France
- Germany (2):
  - GSK Investigational Site, Erlangen
  - GSK Investigational Site, Münster
- Israel (4):
  - GSK Investigational Site, Haifa
  - GSK Investigational Site, Holon
  - GSK Investigational Site, Jerusalem
  - GSK Investigational Site, Rehovot
- Italy (8):
  - GSK Investigational Site, Milan
  - GSK Investigational Site, Modena
  - GSK Investigational Site, Monza
  - GSK Investigational Site, Napoli
  - GSK Investigational Site, Negrar Verona
  - GSK Investigational Site, Padua
  - GSK Investigational Site, Palermo
  - GSK Investigational Site, Roma
- Japan (14):
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Ehime
  - GSK Investigational Site, Fukui
  - GSK Investigational Site, Gunma
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Kagawa
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Nagano
  - GSK Investigational Site, Nagasaki
  - GSK Investigational Site, Nara
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Shizuoka
  - GSK Investigational Site, Tokyo
- Mexico (2):
  - GSK Investigational Site, Mexico City
  - GSK Investigational Site, Monterrey
- Poland (5):
  - GSK Investigational Site, Częstochowa
  - GSK Investigational Site, Katowice
  - GSK Investigational Site, Mysłowice
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Wroclaw
- Russia (3):
  - GSK Investigational Site, Kemerovo
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Samara
- Spain (4):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Valencia
- United Kingdom (10):
  - GSK Investigational Site, Basingstoke
  - GSK Investigational Site, Glasgow
  - GSK Investigational Site, Hull
  - GSK Investigational Site, London
  - GSK Investigational Site, Newcastle upon Tyne
  - GSK Investigational Site, Nottingham
  - GSK Investigational Site, Plymouth
  - GSK Investigational Site, Reading Berkshire
  - GSK Investigational Site, Southampton
  - GSK Investigational Site, Surrey

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com